CLINICAL TRIAL: NCT00907296
Title: A Multi-center, Randomized, Double Blind, Placebo-controlled Study of AMG 785 in Skeletally Mature Adults With a Fresh Unilateral Tibial Diaphyseal Fracture Status Post Definitive Fracture Fixation With an Intramedullary Nail
Brief Title: Study of Romosozumab (AMG 785) in Tibial Diaphyseal Fractures Status Post Intramedullary Nailing
Acronym: STARTT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20062017; 2008-008392-34 (EudraCT Number)
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Results first posted 2019-05-01 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Fracture Healing
Keywords: Fracture Healing; Tibial Diaphyseal Fracture
MeSH Terms: interventions — romosozumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (10):
- Placebo (Placebo Comparator): Participants received subcutaneous injections of matching placebo on day 1 and at weeks 2, 6, and 12.
  Interventions: Drug: Placebo
- Romosozumab 70 mg: 2 Doses (Experimental): Participants received subcutaneous injections of 70 mg romosozumab on day 1 and week 2, and matching placebo at weeks 6 and 12.
  Interventions: Biological: Romosozumab
- Romosozumab 70 mg: 3 Doses (Experimental): Participants received subcutaneous injections of 70 mg romosozumab on day 1 and weeks 2 and 6, and matching placebo at week 12.
  Interventions: Biological: Romosozumab
- Romosozumab 70 mg: 4 Doses (Experimental): Participants received subcutaneous injections of 70 mg romosozumab on day 1 and weeks 2, 6, and 12.
  Interventions: Biological: Romosozumab
- Romosozumab 140 mg: 2 Doses (Experimental): Participants received subcutaneous injections of 140 mg romosozumab on day 1 and week 2, and matching placebo at weeks 6 and 12.
  Interventions: Biological: Romosozumab
- Romosozumab 140 mg: 3 Doses (Experimental): Participants received subcutaneous injections of 140 mg romosozumab on day 1 and weeks 2 and 6, and matching placebo at week 12.
  Interventions: Biological: Romosozumab
- Romosozumab 140 mg: 4 Doses (Experimental): Participants received subcutaneous injections of 140 mg romosozumab on day 1 and weeks 2, 6, and 12.
  Interventions: Biological: Romosozumab
- Romosozumab 210 mg: 2 Doses (Experimental): Participants received subcutaneous injections of 210 mg romosozumab on day 1 and week 2, and matching placebo at weeks 6 and 12.
  Interventions: Biological: Romosozumab
- Romosozumab 210 mg: 3 Doses (Experimental): Participants received subcutaneous injections of 210 mg romosozumab on day 1 and weeks 2 and 6, and matching placebo at week 12.
  Interventions: Biological: Romosozumab
- Romosozumab 210 mg: 4 Doses (Experimental): Participants received subcutaneous injections of 210 mg romosozumab on day 1 and weeks 2, 6, and 12.
  Interventions: Biological: Romosozumab

INTERVENTIONS:
Biological: Romosozumab — Administered by subcutaneous injection
  Other Names: AMG 785; Evenity
  Arms: Romosozumab 140 mg: 2 Doses; Romosozumab 140 mg: 3 Doses; Romosozumab 140 mg: 4 Doses; Romosozumab 210 mg: 2 Doses; Romosozumab 210 mg: 3 Doses; Romosozumab 210 mg: 4 Doses; Romosozumab 70 mg: 2 Doses; Romosozumab 70 mg: 3 Doses; Romosozumab 70 mg: 4 Doses
Drug: Placebo — Administered by subcutaneous injection
  Arms: Placebo

SUMMARY:
The primary objective of this study is to investigate the effect of romosozumab compared with placebo on time to radiographic healing of fresh tibial diaphyseal fractures (fractures in the midsection of the shinbone).

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature adults, age 18 to 85 years with radiographically closed growth plates
* Fresh unilateral closed or Gustilo type I or type II open tibial fracture
* Definitive fracture fixation with reamed (closed and open fractures) or unreamed (open fractures only) intramedullary nailing

Exclusion Criteria:

* Major polytrauma or significant axial trauma
* Associated lower extremity fracture that will delay subject's ability to bear weight beyond the normal time expected for a tibial shaft fracture
* Use of bone grafts at the time of fracture fixation
* Pathological fracture or metabolic or bone disease
* History of symptomatic spinal stenosis or facial nerve paralysis
* Malignancy within the last 5 years
* Evidence of the following (currently or within the past 5 years): elevated transaminases, significantly impaired renal function, current hyper- or hypocalcaemia
* Use of agents affecting bone metabolism
* Subject refuses to use appropriate methods of contraception

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2009-09-02 (Actual); Primary Completion 2012-03-06 (Actual); Study Completion 2013-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (93):
- United States (14):
  - Research Site, Birmingham, Alabama
  - Research Site, Orange, California
  - Research Site, Aurora, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Jacksonville, Florida
  - Research Site, Indianapolis, Indiana
  - Research Site, Detroit, Michigan
  - Research Site, St Louis, Missouri
  - Research Site, Brooklyn, New York
  - Research Site, Rochester, New York
  - Research Site, Altoona, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Columbia, South Carolina
  - Research Site, Sandy City, Utah
- Australia (2):
  - Research Site, Geelong, Victoria
  - Research Site, Parkville, Victoria
- Bulgaria (5):
  - Research Site, Blagoevgrad
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
- Canada (7):
  - Research Site, Red Deer, Alberta
  - Research Site, Ajax, Ontario
  - Research Site, Thunder Bay, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Montreal, Quebec
- Denmark (3):
  - Research Site, Ã…rhus C
  - Research Site, Hvidovre
  - Research Site, KÃ¸benhavn NV
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- France (4):
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Nantes
  - Research Site, Paris
- Germany (5):
  - Research Site, Aachen
  - Research Site, Hamburg
  - Research Site, Hanover
  - Research Site, Mannheim
  - Research Site, Münster
- Greece (4):
  - Research Site, Athens
  - Research Site, Larissa
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, New Territories
- Hungary (4):
  - Research Site, Budapest
  - Research Site, Miskolc
  - Research Site, Nyíregyháza
  - Research Site, Szeged
- India (8):
  - Research Site, Bangalore, Karnataka
  - Research Site, Mangalore, Karnataka
  - Research Site, Pune, Maharashtra
  - Research Site, Jaipur, Rajasthan
  - Research Site, Madurai, Tamil Nadu
  - Research Site, Gandhinagar
  - Research Site, Mangalore
  - Research Site, Nashik
- Italy (5):
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Pisa
  - Research Site, Roma (RM)
  - Research Site, Verona
- Latvia (3):
  - Research Site, Liepāja
  - Research Site, Riga
  - Research Site, Valmiera
- Lithuania (2):
  - Research Site, Kaunas
  - Research Site, Vilnius
- Research Site, Monterrey, Nuevo LeÃ³n, Mexico
- New Zealand (2):
  - Research Site, Christchurch
  - Research Site, Tauranga
- Research Site, Kongsvinger, Norway
- Poland (5):
  - Research Site, Bialystok
  - Research Site, Bytom
  - Research Site, KrakÃ³w
  - Research Site, Krakow
  - Research Site, Lublin
- Romania (2):
  - Research Site, Bucharest
  - Research Site, Timișoara
- Russia (3):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Slovakia (3):
  - Research Site, Bratislava
  - Research Site, Nitra
  - Research Site, Piešťany
- United Kingdom (6):
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Newcastle
  - Research Site, Norwich
  - Research Site, Oxford
  - Research Site, Stanmore

REFERENCES:
- [Background] Bhandari M, Schemitsch EH, Karachalios T, Sancheti P, Poolman RW, Caminis J, Daizadeh N, Dent-Acosta RE, Egbuna O, Chines A, Miclau T. Romosozumab in Skeletally Mature Adults with a Fresh Unilateral Tibial Diaphyseal Fracture: A Randomized Phase-2 Study. J Bone Joint Surg Am. 2020 Aug 19;102(16):1416-1426. doi: 10.2106/JBJS.19.01008. PMID 32358413
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 66 centers in Europe, India, North America, Australia, New Zealand, Hong Kong, and Mexico. Participants were enrolled from 02 September 2009 to 19 September 2011.
Pre-assignment Details: Participants were randomized 1:1:1:1:1:1:1:1:1:3 to 1 of 9 romosozumab treatment groups or placebo. Randomization followed surgery and was stratified by type of fracture and definitive fracture fixation.
Period: Overall Study
Arm/Group | Placebo | Romosozumab 70 mg: 2 Doses | Romosozumab 70 mg: 3 Doses | Romosozumab 70 mg: 4 Doses | Romosozumab 140 mg: 2 Doses | Romosozumab 140 mg: 3 Doses | Romosozumab 140 mg: 4 Doses | Romosozumab 210 mg: 2 Doses | Romosozumab 210 mg: 3 Doses | Romosozumab 210 mg: 4 Doses
Started | 103 | 34 | 34 | 33 | 33 | 33 | 33 | 33 | 31 | 35
Received Treatment | 100 | 34 | 34 | 32 | 33 | 32 | 31 | 32 | 30 | 35
Completed | 83 | 29 | 32 | 29 | 32 | 24 | 27 | 26 | 27 | 28
Not Completed | 20 | 5 | 2 | 4 | 1 | 9 | 6 | 7 | 4 | 7
Not completed — Ineligibility Determined | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Deviation | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Noncompliance | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 7 | 2 | 1 | 1 | 1 | 5 | 3 | 2 | 4 | 2
Not completed — Lost to Follow-up | 9 | 1 | 0 | 2 | 0 | 3 | 2 | 2 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Romosozumab 70 mg: 2 Doses | Romosozumab 70 mg: 3 Doses | Romosozumab 70 mg: 4 Doses | Romosozumab 140 mg: 2 Doses | Romosozumab 140 mg: 3 Doses | Romosozumab 140 mg: 4 Doses | Romosozumab 210 mg: 2 Doses | Romosozumab 210 mg: 3 Doses | Romosozumab 210 mg: 4 Doses | Total
Number analyzed (Participants) | 103 | 34 | 34 | 33 | 33 | 33 | 33 | 33 | 31 | 35 | 402
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (13.8) | 38.6 (13.8) | 43.2 (17.7) | 45.9 (15.6) | 41.3 (13.7) | 41.0 (14.9) | 38.7 (12.7) | 42.8 (13.7) | 36.8 (13.8) | 41.7 (14.4) | 40.9 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 7 | 10 | 8 | 8 | 11 | 11 | 5 | 13 | 12 | 114
  Male | 74 | 27 | 24 | 25 | 25 | 22 | 22 | 28 | 18 | 23 | 288
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 80 | 20 | 24 | 29 | 22 | 23 | 24 | 25 | 24 | 28 | 299
  Black or African American | 2 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 8
  Hispanic or Latino | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 8
  Asian | 20 | 11 | 9 | 3 | 9 | 8 | 8 | 7 | 6 | 5 | 86
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Randomization Stratification [Count of Participants; unit: Participants] — Randomization was stratified according to
  1. Gustilo-Anderson System for classifying open tibial fractures:
     Gustilo type I open fracture: Open tibial fracture with a puncture wound smaller than 1 cm.
     Gustilo type II open fracture: Open tibial fracture with a wound of 1-10 cm.
  2. Definitive fracture fixation: with reamed or unreamed intramedullary (IM) nailing.
  Participants
    Closed with reamed IM nail | 88 | 30 | 30 | 29 | 29 | 29 | 29 | 29 | 28 | 29 | 350
    Gustilo type I/II open with reamed IM nail | 10 | 3 | 4 | 3 | 3 | 4 | 4 | 4 | 3 | 4 | 42
    Gustilo type I/II open with unreamed IM nail | 5 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Time to Radiographic Healing
Description: Time to radiographic healing was defined as the time from intramedullary (IM) nailing to the first occurrence of bridging of 3 out of 4 cortices. Radiographic fracture healing was determined by a panel of independent reviewers (orthopedic/trauma surgeons and radiologists) blinded to treatment.
  The cumulative incidence function (CIF) method was used to estimate the median time to radiographic healing and the confidence intervals. Unplanned revision surgery to promote healing was considered a competing risk in CIF estimate.
Time Frame: 52 weeks
Population: Participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Romosozumab 70 mg: 2 Doses | Romosozumab 70 mg: 3 Doses | Romosozumab 70 mg: 4 Doses | Romosozumab 140 mg: 2 Doses | Romosozumab 140 mg: 3 Doses | Romosozumab 140 mg: 4 Doses | Romosozumab 210 mg: 2 Doses | Romosozumab 210 mg: 3 Doses | Romosozumab 210 mg: 4 Doses
Number analyzed (Participants) | 100 | 34 | 34 | 32 | 33 | 32 | 31 | 32 | 30 | 35
weeks | 16.4 [14.6 to 18.0] | 18.6 [14.0 to 24.4] | 18.3 [13.0 to 21.0] | 18.2 [13.7 to 20.7] | 17.8 [12.6 to 22.9] | 18.1 [13.1 to 20.7] | 17.0 [12.7 to 21.4] | 14.4 [12.6 to 17.0] | 15.4 [13.3 to 17.4] | 16.4 [14.4 to 18.6]
Statistical Analysis 1: Comparison: Placebo vs Romosozumab 70 mg: 2 Doses; The cause-specific hazard was modeled using a Cox proportional hazards model with 10 treatment groups as the independent variable, stratified by type of fracture and definitive fracture fixation (closed with reamed IM nail, Gustilo type I/II open with reamed IM nail, Gustilo type I/II open with unreamed IM nail) and adjusting for quality of surgical fixation; Test type: Superiority; p = 0.3598, Cox proportional hazard model; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.53 to 1.26] — A hazard ratio > 1 favors romosozumab
Statistical Analysis 2: Comparison: Placebo vs Romosozumab 70 mg: 3 Doses; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.6544, Cox proportional hazard model; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.59 to 1.39] — A hazard ratio > 1 favors romosozumab
Statistical Analysis 3: Comparison: Placebo vs Romosozumab 70 mg: 4 Doses; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.9958, Cox proportional hazard model; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.64 to 1.58] — A hazard ratio > 1 favors romosozumab
Statistical Analysis 4: Comparison: Placebo vs Romosozumab 140 mg: 2 Doses; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.6276, Cox proportional hazard model; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.59 to 1.37] — A hazard ratio > 1 favors romosozumab
Statistical Analysis 5: Comparison: Placebo vs Romosozumab 140 mg: 3 Doses; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.8819, Cox proportional hazard model; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.63 to 1.49] — A hazard ratio > 1 favors romosozumab
Statistical Analysis 6: Comparison: Placebo vs Romosozumab 140 mg: 4 Doses; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.7197, Cox proportional hazard model; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.60 to 1.42] — A hazard ratio > 1 favors romosozumab
Statistical Analysis 7: Comparison: Placebo vs Romosozumab 210 mg: 2 Doses; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.6204, Cox proportional hazard model; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.73 to 1.70] — A hazard ratio > 1 favors romosozumab
Statistical Analysis 8: Comparison: Placebo vs Romosozumab 210 mg: 3 Doses; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4779, Cox proportional hazard model; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.75 to 1.84] — A hazard ratio > 1 favors romosozumab
Statistical Analysis 9: Comparison: Placebo vs Romosozumab 210 mg: 4 Doses; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.9952, Cox proportional hazard model; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.65 to 1.53] — A hazard ratio > 1 favors romosozumab

2. Secondary Outcome: Change From Week 8 in Short Form (36) Health Survey Physical Functioning Domain
Description: The Medical Outcome Study Short Form 36-Item Health Survey (SF-36), Version 2, is a self-administered instrument that measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). The physical functioning domain includes 10 questions that assess limitations in physical activities because of health problems.
  Norm-based scores were used in analyses, calibrated so that 50 is the average score and the standard deviation equals 10. The range of SF-36 physical functioning is 14.94 - 57.03. Higher scores indicate a higher level of functioning. A positive change from baseline score indicates an improvement in physical functioning.
Time Frame: Week 8 and weeks 12, 16, 20, 24, 36, and 52
Population: Participants who received at least 1 dose of study drug and with available data at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Romosozumab 70 mg: 2 Doses | Romosozumab 70 mg: 3 Doses | Romosozumab 70 mg: 4 Doses | Romosozumab 140 mg: 2 Doses | Romosozumab 140 mg: 3 Doses | Romosozumab 140 mg: 4 Doses | Romosozumab 210 mg: 2 Doses | Romosozumab 210 mg: 3 Doses | Romosozumab 210 mg: 4 Doses
Number analyzed (Participants) | 100 | 34 | 34 | 32 | 33 | 32 | 31 | 32 | 30 | 35
units on a scale
  Week 12: number analyzed (Participants) | 88 | 26 | 28 | 28 | 29 | 29 | 24 | 27 | 27 | 30
  Week 12 | 5.77 (9.90) | 6.31 (6.84) | 5.67 (8.60) | 5.04 (9.01) | 4.28 (8.22) | 7.08 (8.06) | 3.63 (9.30) | 3.65 (9.06) | 7.33 (7.99) | 5.64 (6.67)
  Week 16: number analyzed (Participants) | 85 | 24 | 27 | 27 | 28 | 29 | 23 | 28 | 25 | 28
  Week 16 | 9.64 (10.36) | 9.83 (7.24) | 9.19 (11.30) | 9.28 (11.14) | 8.89 (10.71) | 11.18 (9.23) | 8.78 (11.34) | 9.23 (9.59) | 9.50 (9.01) | 9.01 (10.41)
  Week 20: number analyzed (Participants) | 83 | 21 | 25 | 26 | 30 | 27 | 22 | 25 | 24 | 25
  Week 20 | 13.20 (12.25) | 14.53 (9.69) | 10.45 (11.66) | 13.50 (12.02) | 12.13 (10.88) | 14.77 (13.52) | 12.44 (11.97) | 12.61 (10.88) | 12.50 (10.76) | 11.05 (11.56)
  Week 24: number analyzed (Participants) | 80 | 25 | 24 | 27 | 28 | 24 | 20 | 25 | 24 | 26
  Week 24 | 15.87 (11.55) | 15.07 (9.31) | 10.34 (13.31) | 15.90 (11.26) | 14.57 (10.34) | 16.84 (12.70) | 11.79 (17.64) | 13.05 (10.99) | 13.05 (10.25) | 12.38 (14.04)
  Week 36: number analyzed (Participants) | 79 | 25 | 25 | 27 | 27 | 26 | 24 | 23 | 26 | 26
  Week 36 | 19.57 (11.60) | 20.96 (11.68) | 11.48 (17.84) | 17.23 (10.15) | 17.61 (11.03) | 19.43 (12.83) | 15.70 (19.03) | 15.01 (11.23) | 17.47 (14.34) | 15.22 (15.20)
  Week 52: number analyzed (Participants) | 78 | 26 | 27 | 26 | 30 | 23 | 24 | 24 | 26 | 26
  Week 52 | 20.74 (11.96) | 23.47 (11.55) | 13.63 (19.04) | 19.02 (10.80) | 19.63 (12.17) | 24.80 (11.24) | 17.19 (15.51) | 15.50 (13.17) | 18.29 (14.94) | 15.44 (17.15)

3. Secondary Outcome: Number of Participants With Unplanned Revision Surgeries
Time Frame: 52 weeks
Population: Participants who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Romosozumab 70 mg: 2 Doses | Romosozumab 70 mg: 3 Doses | Romosozumab 70 mg: 4 Doses | Romosozumab 140 mg: 2 Doses | Romosozumab 140 mg: 3 Doses | Romosozumab 140 mg: 4 Doses | Romosozumab 210 mg: 2 Doses | Romosozumab 210 mg: 3 Doses | Romosozumab 210 mg: 4 Doses
Number analyzed (Participants) | 100 | 34 | 34 | 32 | 33 | 32 | 31 | 32 | 30 | 35
Participants | 8 | 1 | 3 | 3 | 1 | 0 | 0 | 0 | 1 | 1

4. Secondary Outcome: Time to Clinical Healing
Description: Time to clinical healing was defined as the time from the IM nailing surgery date to the first date that both the score for ability to bear weight on the fractured limb and the score for absence of pain at the fracture site were equal to 6.
  The score for the ability to bear weight on the fractured limb was based on the ability to stand on affected leg without assistive device and the ability to walk without assistive device. The score ranges from 0 (unable to bear full body weight on the fractured limb) to 6 (able to bear full body weight on the fractured limb). Absence of pain at the fracture site was based on the absence of pain at the fracture site when applying direct pressure to the fracture site and applying a stress to the fracture site. The score ranges from 0 (pain without palpation at fracture site) to 6 (total absence of pain at fracture site).
  Time to clinical healing was estimated using CIF; unplanned revision surgery was considered a competing risk in CIF estimate.
Time Frame: 52 weeks
Population: Participants who received at least 1 dose of study drug
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Romosozumab 70 mg: 2 Doses | Romosozumab 70 mg: 3 Doses | Romosozumab 70 mg: 4 Doses | Romosozumab 140 mg: 2 Doses | Romosozumab 140 mg: 3 Doses | Romosozumab 140 mg: 4 Doses | Romosozumab 210 mg: 2 Doses | Romosozumab 210 mg: 3 Doses | Romosozumab 210 mg: 4 Doses
Number analyzed (Participants) | 100 | 34 | 34 | 32 | 33 | 32 | 31 | 32 | 30 | 35
weeks | 18.4 [16.6 to 20.4] | 21.4 [15.7 to 28.6] | 18.3 [14.4 to 22.4] | 17.1 [14.4 to 21.0] | 20.8 [12.6 to 28.0] | 22.3 [15.0 to 24.3] | 15.0 [12.6 to 17.0] | 16.3 [12.4 to 21.0] | 14.6 [12.9 to 18.6] | 17.6 [14.9 to 19.7]
Statistical Analysis 1: Comparison: Placebo vs Romosozumab 70 mg: 2 Doses; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1713, Cox proportional hazard model; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.47 to 1.14] — A hazard ratio > 1 favors romosozumab
Statistical Analysis 2: Comparison: Placebo vs Romosozumab 70 mg: 3 Doses; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.9958, Cox proportional hazard model; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.65 to 1.53] — A hazard ratio > 1 favors romosozumab
Statistical Analysis 3: Comparison: Placebo vs Romosozumab 70 mg: 4 Doses; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.2950, Cox proportional hazard model; Hazard Ratio (HR) = 1.27, 95% CI 2-sided [0.81 to 1.97] — A hazard ratio > 1 favors romosozumab
Statistical Analysis 4: Comparison: Placebo vs Romosozumab 140 mg: 2 Doses; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0844, Cox proportional hazard model; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.44 to 1.05] — A hazard ratio > 1 favors romosozumab
Statistical Analysis 5: Comparison: Placebo vs Romosozumab 140 mg: 3 Doses; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.3225, Cox proportional hazard model; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.52 to 1.24] — A hazard ratio > 1 favors romosozumab
Statistical Analysis 6: Comparison: Placebo vs Romosozumab 140 mg: 4 Doses; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.4754, Cox proportional hazard model; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [0.76 to 1.81] — A hazard ratio > 1 favors romosozumab
Statistical Analysis 7: Comparison: Placebo vs Romosozumab 210 mg: 2 Doses; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.5578, Cox proportional hazard model; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.74 to 1.75] — A hazard ratio > 1 favors romosozumab
Statistical Analysis 8: Comparison: Placebo vs Romosozumab 210 mg: 3 Doses; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1864, Cox proportional hazard model; Hazard Ratio (HR) = 1.34, 95% CI 2-sided [0.87 to 2.07] — A hazard ratio > 1 favors romosozumab
Statistical Analysis 9: Comparison: Placebo vs Romosozumab 210 mg: 4 Doses; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.8488, Cox proportional hazard model; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.68 to 1.59] — A hazard ratio > 1 favors romosozumab

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Placebo | Romosozumab 70 mg: 2 Doses | Romosozumab 70 mg: 3 Doses | Romosozumab 70 mg: 4 Doses | Romosozumab 140 mg: 2 Doses | Romosozumab 140 mg: 3 Doses | Romosozumab 140 mg: 4 Doses | Romosozumab 210 mg: 2 Doses | Romosozumab 210 mg: 3 Doses | Romosozumab 210 mg: 4 Doses
Serious Adverse Events (participants affected / at risk) | 10/100 | 4/34 | 2/34 | 3/32 | 3/33 | 4/32 | 2/31 | 3/32 | 3/30 | 0/35
Other Adverse Events (participants affected / at risk) | 38/100 | 9/34 | 17/34 | 12/32 | 16/33 | 7/32 | 9/31 | 10/32 | 9/30 | 6/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=100) | Romosozumab 70 mg: 2 Doses (N=34) | Romosozumab 70 mg: 3 Doses (N=34) | Romosozumab 70 mg: 4 Doses (N=32) | Romosozumab 140 mg: 2 Doses (N=33) | Romosozumab 140 mg: 3 Doses (N=32) | Romosozumab 140 mg: 4 Doses (N=31) | Romosozumab 210 mg: 2 Doses (N=32) | Romosozumab 210 mg: 3 Doses (N=30) | Romosozumab 210 mg: 4 Doses (N=35)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device breakage (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Bone fissure (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Loss of anatomical alignment after fracture reduction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paraplegia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Medical device removal (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular insufficiency (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=100) | Romosozumab 70 mg: 2 Doses (N=34) | Romosozumab 70 mg: 3 Doses (N=34) | Romosozumab 70 mg: 4 Doses (N=32) | Romosozumab 140 mg: 2 Doses (N=33) | Romosozumab 140 mg: 3 Doses (N=32) | Romosozumab 140 mg: 4 Doses (N=31) | Romosozumab 210 mg: 2 Doses (N=32) | Romosozumab 210 mg: 3 Doses (N=30) | Romosozumab 210 mg: 4 Doses (N=35)
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 2 | 0 | 0 | 1 | 3 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Medical device discomfort (General disorders) | 3 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 6 | 0 | 4 | 4 | 3 | 2 | 1 | 3 | 2 | 1
Pain (General disorders) | 7 | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 5 | 2 | 1 | 0 | 0 | 2 | 1 | 2 | 1 | 1
Influenza (Infections and infestations) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 4 | 2 | 2 | 0 | 2 | 0 | 0 | 1 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 4 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 1 | 1 | 5 | 4 | 3 | 0 | 4 | 2 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 3 | 1 | 1 | 0 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 0 | 0 | 0 | 1 | 2 | 3 | 1 | 1 | 0
Headache (Nervous system disorders) | 3 | 0 | 2 | 0 | 0 | 1 | 2 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 5 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.